CLINICAL TRIAL: NCT06758882
Title: Surgical Treatment With or Without Apalutamide in Subjects With High Risk Prostate Cancer Who Are Candidates for Radical Prostatectomy and Staged as Oligometastatic With PSMA-PET
Acronym: STAPLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marco Oderda (Other)
Responsible Party: Sponsor-Investigator, Marco Oderda, Principal Investigator, A.O.U. Città della Salute e della Scienza
Organization: A.O.U. Città della Salute e della Scienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40/2023; 2022-002844-37 (EudraCT Number)
Record Dates: First submitted 2024-11-19; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: High Risk Prostate Cancer
Keywords: oligometastatic at PSMA PET/CT; apalutamide; radical prostatectomy; pelvic lymph node dissection; androgen deprivation therapy (ADT)
MeSH Terms: interventions — apalutamide; Receptors, Androgen

STUDY DESIGN:
Intervention Model Description: randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Experimental): radical prostatectomy + apalutamide + androgen deprivation therapy
  Interventions: Drug: Apalutamide; Drug: Androgen receptor (AR) inhibitor
- Control Group (Active Comparator): radical prostatectomy + androgen deprivation therapy
  Interventions: Drug: Androgen receptor (AR) inhibitor

INTERVENTIONS:
Drug: Apalutamide — administration of non steroid androgenic receptor inhibitors plus androgen deprivation therapy
  Arms: Interventional Group
Drug: Androgen receptor (AR) inhibitor — administration of androgen deprivation therapy

SUMMARY:
This is a phase 2, open-label, randomized study of adjuvant treatment in subjects with high-risk prostate cancer who are candidates for RP with PLND based on M0 status at conventional imaging, but staged as oligometastatic with PSMA PET/CT (performed as routine practice, according to recent evidence on high-risk prostate cancer patients). Ninety-four subjects will receive apalutamide plus ADT or ADT alone after surgery. ADT is defined as medical castration (ie, gonadotropin-releasing hormone analogues [GnRHa, agonist or antagonist]). Subjects will be randomly assigned in a 1:1 ratio to receive apalutamide plus ADT or ADT alone.

Patients randomized to receive ADT + apalutamide or ADT alone will begin their adjuvant treatment 4 weeks (28 to 32 days) after surgery. A first dosage of PSA and testosterone will be performed just before starting adjuvant therapy but not before 28 days from surgery. Subsequently, PSA and testosterone dosage and clinical visits will be performed after 3 months from surgery and every 3 months until completion of study. PSMA PET/CT scan will be performed yearly, or in case of PSA progression. The Posttreatment Follow-up Phase will begin after 18 months of ADT and will last for 6 months, until study completion. Afterwards, patients will continue their follow-up according to the best clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age, < 80 years of age
2. Signed informed consent form (ICF) indicating that the subject understands the purpose and procedures required for the study and is willing to participate in the study; subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol (Section 4.3)
3. Histologically confirmed adenocarcinoma of the prostate
4. High-risk disease defined by a total Gleason Sum Score ≥ 4+4 (=Grade Groups [GG] 4-5)
5. Conventional imaging negative for metastases
6. Presence of low volume metastatic disease at pre-surgery PSMA PET/CT. The metastatic burden is classified according to the definition used in the CHARTEED trial applied to PSMA PET/CT, where high metastatic burden was defined as four or more bone metastases with one or more outside the vertebral bodies or pelvis, or visceral metastases, or both; all other assessable patients were considered to have low metastatic burden
7. Candidate to RP with PLND
8. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
9. Adequate organ function determined by the following laboratory values:

   1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin within normal limits, ie, ≤ the upper limit of normal [ULN] (note that in subjects with Gilbert's syndrome, if total bilirubin is >1.5 X ULN, measure direct and indirect bilirubin. If direct bilirubin is ≤1.5 X ULN, the subject may be eligible);
   2. Serum creatinine <1.8 mg/dL;
   3. Platelets ≥75.000/dL, without transfusion and/or growth factors within 56 days prior to RP;
   4. Haemoglobin ≥11.0 g/dL, without transfusion and/or growth factors within 56 days prior to RP;
10. Able to receive ADT for at least 18 months, based on cardiovascular risk assessment and the investigator's assessment
11. Be able to swallow whole study drug tablets

Exclusion Criteria:

1. Distant metastasis based on conventional imaging (CT scan or bone scintigraphy). Nodal disease below the iliac bifurcation (clinical stage N1 at CT scan) is not an exclusion criterion.
2. Prior hormonal treatment (GnRHa, agonist or antagonist)
3. Prior bilateral orchiectomy
4. History of prior systemic or local therapy for prostate cancer, including pelvic radiation and whole gland or focal ablative modalities for prostate cancer
5. Use of any investigational agent ≤4 weeks prior to RP or any therapeutic procedure for prostate cancer at any time
6. Major surgery ≤4 weeks prior to RP
7. Any of the following within 12 months prior to first dose of study drug: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias or New York Heart Association Class II to IV heart disease; uncomplicated deep vein thrombosis is not considered exclusionary
8. Human immunodeficiency virus-positive subjects with 1 or more of the following: (1) not receiving highly active antiretroviral therapy; (2) had a change in antiretroviral therapy within 6 months of the start of screening; (3) receiving antiretroviral therapy that may interfere with study drug (consult Sponsor for review of medication prior to enrolment); (4) CD4 count <350 at screening; (5) AIDS-defining opportunistic infection within 6 months of start of screening; (6) active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction
9. History of seizure; any condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness ≤1 year prior to RP); presence of brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect
10. Patients taking any prohibited medications (as reported in session 6.2 of the protocol, including medicinal products known to prolong the QT interval and/or drugs commonly known to cause torsade de pointes and/or drugs known to lower the seizure threshold within 4 weeks prior to RP) should not be included
11. Gastrointestinal conditions affecting absorption
12. Known or suspected contraindications or hypersensitivity to apalutamide, GnRHa or any of the components of the formulations
13. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject
14. Active malignancies (ie, progressing or requiring treatment or treatment change in the last 24 months) other than prostate cancer. The only allowed exceptions are: non-muscle invasive bladder cancer (NMIBC); skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured; breast cancer (adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence); malignancy that is considered cured with minimal risk of recurrence.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Radiological progression-free survival (RPFS) | from date of randomization to 24 months (6 months of follow-up after 18 months of treatment)
  the time from randomization to date of first PSMA PET/CT-based documentation of progressive disease (appearance of new lesions) or death, whichever occurred first. The RECIP criteria for progression will also be used for the analysis.

SECONDARY OUTCOMES:
Adverse events (AEs) | from date of randomization to 24 months (6 months of follow-up after 18 months of treatment)
  Adverse events (AEs) will be graded according to the CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Surgical Sciences - Urology, Molinette Hospital, University of Torino, Torino, To, Italy